CLINICAL TRIAL: NCT05460351
Title: Effect of Beetroot Juice on Body Composition, Physical Function, Muscle Strength, and Peak Oxygen Consumption in Resistance Trained Older Adults Consuming a Protein Supplement
Brief Title: Beetroot Juice Resistance Training Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Principal Investigator, Gary Miller, Professor, Wake Forest University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00025941
Record Dates: First submitted 2022-07-04; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Sarcopenia; Old Age; Atrophy
MeSH Terms: conditions — Sarcopenia; Atrophy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups. The first group will consume daily beetroot juice containing 380 mg of nitrate and the second group will consume daily beetroot juice with nitrate removed. Both groups will undergo resistance exercise training and consume a protein supplement
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A third party not involved with the conduct of the study provided research staff with the beetroot juice in participant specific coded bottles. The research staff then distributed these coded bottles to the participant. At the end of the trial, the code was revealed for intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRJ+Nitrate (Experimental): This arm underwent a 3 days a week, 10 weeks of resistance exercise training program and consumed for a 70 mL bottle of beetroot juice containing 380 mg of nitrate plus a 15 dose of whey protein after each exercise session.
  Interventions: Dietary Supplement: BRJ+Nitrate
- Control (Placebo Comparator): This arm underwent a 3 days a week, 10 weeks of resistance exercise training program and consumed for a 70 mL bottle of beetroot juice containing 0 mg of nitrate plus a 15 dose of whey protein after each exercise session.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: BRJ+Nitrate — Participants in this group drank a 70 mL bottle of Beet It Sport drink with nitrate plus 15 grams of whey protein 3 days a week following a resistance exercise training program
  Arms: BRJ+Nitrate
Dietary Supplement: Control — Participants in this group drank a 70 mL bottle of Beet It Sport drink without nitrate plus 15 grams of whey protein 3 days a week following a resistance exercise training program
  Arms: Control

SUMMARY:
The present study compared the effects of a nitrate containing beetroot juice supplement (BRJ+Nitrate) vs. a placebo (Control) on total and regional fat free mass, quadriceps muscle strength, lower body mobility, and VO2peak in healthy, older adults undergoing a 10-week long progressive resistance training program with protein supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide own transportation to study testing visits and intervention
* Able to read and write in English
* Nondiabetic, i.e. fasting glucose < 126 mg/dl
* Sedentary (less than 60 minutes of moderate intensity structured physical activity each week and occurs in no more than 10 minute blocks and not participating in a resistance exercise training program)
* Willingness to provide informed consent and participate in intervention. Participants with diagnosed depression were permitted to participate provided that they have been medically stable without medication change for at least 3 months.

Exclusion Criteria:

* Smoking or use of chewing tobacco
* Involved in another intervention research study
* Diabetic (type 1 or 2)
* Atrophic gastritis
* Hypo- or hyperthyroidism
* Gout or history of kidney stones
* History of hypotension
* Premenopausal (women)
* Aversion to study-related testing procedures
* Allergy/sensitivity/aversion to beetroot beverages or protein supplement
* Medical conditions with contraindications for engaging in resistance training program or taking the protein supplement
* Systemic, uncontrolled diseases (diabetes, recent (last 6 months) or current treatment of cancer, thyroid disorders, cardiovascular disease, COPD, or inflammatory bowel diseases)
* Use of any of the following medications: phosphodiesterase type 5 inhibitors, nitroglycerin or nitrate preparations, proton pump inhibitors, or medications for hypothyroidism
* Potential inability to complete the tasks required for the protocol as well as conditions that may interfere with interpretation of results including: inability to ambulate, severe congestive heart failure or severe cardiovascular disease, neoplasm for practical and neurophysiologic reasons
* Individuals with contraindications for performing a graded exercise test or have medical contraindications for participating in a scheduled exercise training program
* Individuals more than 300 pounds or less than 125 pounds due to DEXA weight limits and possibility of exceeding recommended daily nitrate dose of 7 mg/kg body weight, respectively.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Whole body fat free mass | Collected at baseline
  Mass of fat free tissue
Whole body fat mass | Collected at baseline
  Mass of fat tissue
Thigh muscle | Collected at baseline
  Volume of thigh muscle
Thigh intermuscular fat | Collected at baseline
  Volume of fat in the thigh muscle
Thigh subcutaneous fat | Collected at baseline
  Volume of subcutaneous fat in the thigh
Visceral fat | Collected at baseline
  Volume of visceral fat
Muscle strength | Collected at baseline
  Strength of quadriceps muscle at a speed of 60 degrees per second
400 meter walk | Collected at baseline
  Time to walk 400 meters
Stair climb time | Collected at baseline
  Time to ascend and descend 12 stairs
Peak oxygen consumption | Collected at baseline
  Peak oxygen consumed at maximal exercise during graded exercise testing
Whole body fat free mass | Collected at 10-weeks
  mass of fat free tissue
Whole body fat mass | Collected at 10-weeks
  Mass of fat tissue
Thigh muscle | Collected at 10-weeks
  Volume of thigh muscle
Thigh intermuscular fat | Collected at 10-weeks
  Volume of fat in the thigh muscle
Thigh subcutaneous fat | Collected at 10-weeks
  Volume of subcutaneous fat in the thigh
Visceral fat | Collected at 10-weeks
  Volume of visceral fat
Muscle strength | Collected at 10-weeks
  Strength of quadriceps muscle at a speed of 60 degrees per second
400 meter walk | Collected at 10-weeks
  Time to walk 400 meters
Stair climb time | Collected at 10-weeks
  Time to ascend and descend 12 stairs

IPD SHARING:
Plan to Share IPD: No